CLINICAL TRIAL: NCT06659653
Title: Safety and Effectiveness of PRG2302 (CD19/CD22-targeting CAR-T Cells) for Refractory or Relapsed B-cell Acute Lymphoblastic Leukemia Disease.
Brief Title: Safety and Efficacy of PRG-2302 for Refractory or Relapsed B-cell Acute Lymphoblastic Leukemia Disease.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tan Jie (Other)
Collaborators: Shenzhen Pregene Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Tan Jie, Professor, The First People's Hospital of Jingzhou
Organization: The First People's Hospital of Jingzhou (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG2302
Record Dates: First submitted 2024-09-05; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CAR-T
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment (Experimental): Plan to design three dose levels (0.5x10^6 CAR-T/kg ，1.0x10^6 CAR-T/kg and 2.0x10^6 CAR-T/kg ), with 3-6 R/R B-ALL subjects included in each dose group, totaling 9-18 subjects. Within each dose group, the next subject can be administered after the previous subject has completed at least 14 days of safety observation.
  Interventions: Drug: PRG2302

INTERVENTIONS:
Drug: PRG2302 — Dose group 1: with a dosage of 0.5x10^6 (cells/kg) per dose Dose group 2: with a dosage of 1.0x10^6 (cells/kg) per dose Dose group 3: with a dosage of 2.0x10^6 (cells/kg) per dose

SUMMARY:
A Clinical Study on the Safety and Effectiveness of CD19/CD22 Chimeric Antigen Receptor T Cells in the Treatment of Refractory or Relapsed B-cell Acute Lymphoblastic Leukemia Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, not over 70 years old (including 70 years old);
2. Meet the following diagnostic criteria for recurrent or refractory B-ALL:

A clear diagnosis of B-cell acute lymphoblastic leukemia with any of the following conditions Patients:

* recurrent: recurrence within 12 months after the first remission after standard treatment;
* refractory:

  1.induction No remission after more than 6 weeks of treatment or two courses of induction therapy; 2.Two or more CR or CRIs Later recurrence; 3.Relapse for the first time after chemotherapy and no remission after at least one salvage treatment; 4.Recurrence after autologous or allogeneic hematopoietic stem cell transplantation;

  3. Bone marrow or peripheral blood flow cytometry showed positive CD19 and/or CD22 leukemia cells;

  4.The proportion of primitive and naive lymphocyte in bone marrow during screening period was ≥ 5%;

  5.The functions of important organs are basically normal:
  1. Echocardiography indicated cardiac ejection fraction ≥50%, and no obvious abnormality was found in electrocardiogram;
  2. Renal function: creatinine clearance (CrCl) (Cockcroft-Gault formula, Appendix 4) ≥30mL/min;
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0× upper limit of normal value (ULN);
  4. Total bilirubin (TBIL) and alkaline phosphatase (AKP or ALP)

     * 2.0×ULN (Gilbert syndrome ≤ 3.0×ULN);
  5. Blood oxygen saturation >92%;
  6. Expected survival≥3 months;
  7. ECOG score : 0~2;
  8. Willing and signed informed consent.

     Exclusion Criteria:

  <!-- -->

  1. Active central nervous system (CNS) leukemia (NCCN guidelines defined as CNS-3 grade and CNS-2 patients with neurological symptoms);
  2. Subjects with other malignancies within 5 years (except patients who have been cured and have no active disease for more than 3 years prior to screening, and patients with non-melanoma skin cancer, basal cell or squamous cell skin cancer, local prostate cancer, ductal carcinoma in situ, papillary or follicular thyroid cancer, and carcinoma in situ);
  3. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive and peripheral blood hepatitis B virus (HBV) DNA titer greater than the normal range; Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA titer greater than the normal range; Positive for human immunodeficiency virus (HIV) antibodies; Syphilis positive; Peripheral blood tests positive for cytomegalovirus (CMV) and/or Epstein-Barr virus (EBV);
  4. There is an uncontrolled active infection;
  5. Patients with clinically significant diseases of the central nervous system, such as epilepsy, cerebrovascular ischemia/bleeding history, cerebellar diseases or other organic brain syndromes or psychosis (except those with previous central invasion but improved after treatment);
  6. Organ failure patients:

  <!-- -->

  1. Heart:

     a.New York Heart Association (NYHA) Stage III or IV congestive heart failure; b.Had a myocardial infarction or received coronary artery bypass grafting (CABG) or coronary stenting within 6 months or less before signing the ICF; c.A history of clinically significant ventricular arrhythmia, or unexplained syncope (other than those due to vasovagal or dehydration); d.History of severe non-ischemic cardiomyopathy;
  2. Liver:

     According to the Wuhan Conference Classification (1983) to reach level III or above;
  3. kidney: Renal insufficiency reaches stage III renal failure or above;

  7.Any serious and/or uncontrollable comorbidities that the investigator believes may interfere with the assessment during the study;

  8.Known allergic reactions, hypersensitivities, intolerances, or contraindications to any component of PRG2302 or the drugs that may be used in the study (including fludarabine, cyclophosphamide, tolumab, albumin), or prior severe allergic reactions;

  9.Donor lymphocyte infusion (DLI) was received within 4 weeks prior to anapheresis.

  10.Live/attenuated vaccine was administered within 4 weeks prior to anapheresis or during the planned study period;

  11.Major surgery or surgical treatment within 4 weeks for any reason;

  12.Patients with a history of allogeneic hematopoietic stem cell transplantation in the 4 weeks prior to the collection, acute graft-versus-host disease (GvHD) or moderate-to-severe chronic grade 2 to 4 GvHD in the 4 weeks prior to collection, requiring systemic drug therapy (such as hormones or other immunosuppressants);

  13.High doses of chemotherapy within 2 to 4 weeks, intrathecal therapy within 1 week, short-acting cytotoxic drugs, TKI and systemic glucocorticoid therapy within 3 days, or biologic drugs for disease treatment within 4 weeks;

  14.Pregnant women and breastfeeding women cannot stop breastfeeding, and fertile men and their partners or women refuse to use effective contraceptive methods during the study period and at the end of the study (1 year after transfusion);In the researchers' judgment, a patient is fertile: he/she is biologically capable of having children and having a normal sexual life.Female patients who are infertile (i.e. meet at least 1 of the following criteria) : Have undergone hysterectomy or bilateral oophorectomy or bilateral tubal ligation, or have medically confirmed ovarian failure, or have medically confirmed postmenopause (at least 12 consecutive months of menopause);

  15.Patients who cannot collect a sufficient number of mononuclear cells or T cells (e.g., failure to establish a collection pathway, collection failure, or low T cell proportion during screening);

  16.Participated in other intervention clinical trials within 3 months;

  17.Other medical conditions determined by the investigator to be unsuitable for lymphocyte clearance or cell infusion or other unsuitable participants for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Safe dose of PRG-2302 infusion | Up to 24 months after PRG-2302 infusion
  To evaluate the safe dose of PRG-2302 infusion, 3 dosage group were designed in this trial, they are 0.5×10^6 CAR-T,1.0×10^6 CAR-T, and 2.0×10^6 CAR-T
Occurrence of AE after PRG-2302 infusion | Up to 24 months after PRG-2302 infusion
  To evaluate the occurrence of AE after PRG-2302 infusion based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Jingzhou, Jinzhou, Hubei, China

IPD SHARING:
Plan to Share IPD: No